CLINICAL TRIAL: NCT02279511
Title: Evaluating the Effectiveness of the Use of Intravenous Infusions of Adenosine Triphosphate (ATP) in Patients With Moderate Alzheimer's Disease and Severe: Double-blind Dose Finding Clinical Trial.
Brief Title: ATP in Alzheimer Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sara Varea (Other)
Responsible Party: Sponsor-Investigator, Sara Varea, Clinical Trial Manager, Fundacion Clinic per a la Recerca Biomédica
Organization: Fundacion Clinic per a la Recerca Biomédica (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: ECA4A
Record Dates: First submitted 2014-10-22; First posted 2014-10-31 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer
MeSH Terms: conditions — Alzheimer Disease | interventions — Adenosine Triphosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 24 hours infusion of ATP (Experimental)
  Interventions: Drug: ADENOSINE TRIPHOSPHATE
- 6 hours infusion of ATP (Experimental)
  Interventions: Drug: ADENOSINE TRIPHOSPHATE
- 24 hours infusion of placebo (Placebo Comparator)
  Interventions: Drug: PLACEBO
- 6 hours infusion of placebo (Placebo Comparator)
  Interventions: Drug: PLACEBO

INTERVENTIONS:
Drug: ADENOSINE TRIPHOSPHATE — Infusion of 2.5g of ATP in 500 mL of saline solution. (IV)
  Other Names: ATP
  Arms: 24 hours infusion of ATP; 6 hours infusion of ATP
Drug: PLACEBO — Infusion of 500 mL of saline solution. (IV)
  Arms: 24 hours infusion of placebo; 6 hours infusion of placebo

SUMMARY:
To Check whether systemic treatment with ATP alters the profile of cerebral metabolism in patients with Alzheimer's disease using MRS techniques (Magnetic Resonance Spectroscopy) and adjust the infusion (minimum effective dose) that promotes this metabolic change.

ELIGIBILITY:
Inclusion Criteria:

* 1. Men and women aged 55-85 years
* 2. Diagnosis of possible or probable Alzheimer disease according to NIA-AA 2011 criteria.
* 3. Global Deterioration Scale Stadium 5-6 / 15-5 Mini-mental State examination
* 4. The patient is living with a family as a primary caregiver or a caregiver trained to accompany adequate and all intervention and follow-up visits. Patient and caregiver knowledge of local languages sufficient.
* 5. The patient and caregiver willing to participate in the study. There is a high probability that patient and caregiver to complete the study.
* 6. The patient has no sensory deficits preventing evaluation.
* 7. The patient receives a stable Alzheimer Disease conventional medication. No change in treatment at least 90 days prior to selection.
* 8. The patient receives a conventional stable medication for possible comorbidities. No change in treatment at least 90 days prior to selection.
* 9. The subject or his legal representative give prior informed consent that includes genetic studies of Apolipoprotein E and rs11870474.

Exclusion Criteria:

* 1. Concomitant severe neurological disease Alzheimer Disease.
* 2. Presence or history of psychiatric disorders with an emphasis on positive behavioral disorders associated with Alzheimer Disease (aggressiveness, agitation, delusions, hallucinations, anxiety).
* 3. Current Severe systemic disease that may prevent completion of the study.
* 4. History STROKE.
* 5. History of convulsions and use of anticonvulsants.
* 6. History of myocardial infarction, angina pectoris, cardiac arrhythmias and other serious cardiovascular disorders such as congestive heart failure, and valvular aneurysms.
* 7. Background Diabetes mellitus and / or pictures of hypoglycemia.
* 8. Uncontrolled hypertension (systolic> 160 mmHg and / or Diastolic> 95 mmHg).
* 9. Systemic hypotension (SBP <86 mmHg) or bradycardia (<50 beats per minute)
* 10. Bronchial Asthma History or lung diseases that cause bronchospasm or bronchoconstriction
* 11. Kidney failure (patients with medical restrictions or income parenteral intake of fluids).
* 12. Liver failure.
* 13. Respiratory failure (need supplemental oxygen supply)
* 14. Blood donation in the last 90 days or anemia (Hb <10g/dL)
* 15. Use connection (<30 days prior to screening) of antidepressants, sedatives and hypnotics.
* 16. Using Alzheimer Disease experimental drugs in the last 60 days prior to screening.
* 17. Women who are pregnant or fertile
* 18. Inadequate venous access to prevent parenteral administration of infusions.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Detection of brain metabolic changes after ATP infusion by spectroscopy techniques (H + MRS) | expected average of 7-25 hours post infusion
  Spectroscopy will be taken one hour after the infusion (7h for patients allocated to 6h arm and 25h in 24h infusion arm)
Changes in Cogstate results | expected average of 7-25 hours post infusion
  one hour after the infusion (7h for patients allocated to 6h arm and 25h in 24h infusion arm)

SECONDARY OUTCOMES:
Changes in Cogstate results | 3 months compared to baseline.
  The cogstate is a software used to evaluate cognitive impairment
Changes in test Mini-Mental State Examination | 3 months compared to baseline.
Changes in synaptic activity after treatment administration Neurological examination | post treatment or 3 months post baseline
Electrocardiogram results | an expected average of 90 days
adverse events | at 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Mercè Boada Rovira, MD PhD, Principal Investigator — Fundació ACE. Barcelona Alzheimer Treatment and Research Center
Locations (2):
- Spain (2):
  - Fundació ACE, Barcelona, Barcelona
  - Hospital Sanitas CIMA, Barcelona